CLINICAL TRIAL: NCT07229118
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered COR-1004
Brief Title: A Study to Evaluate COR-1004 in Adult Volunteers.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corsera Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: COR-PCS-25-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; lipid-lowering therapy
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 - Dose 1 of COR-1004 (Experimental): A single dose of COR-1004 will be administered subcutaneously
  Interventions: Drug: COR-1004
- Cohort 1 - Placebo (Placebo Comparator): A single dose of placebo will be administered subcutaneously
  Interventions: Drug: Placebo
- Cohort 2 - Dose 2 of COR-1004 (Experimental): A single dose of COR-1004 will be administered subcutaneously
  Interventions: Drug: COR-1004
- Cohort 2 - Placebo (Placebo Comparator): A single dose of placebo will be administered subcutaneously
  Interventions: Drug: Placebo
- Cohort 3 - Dose 3 of COR-1004 (Experimental): A single dose of COR-1004 will be administered subcutaneously
  Interventions: Drug: COR-1004
- Cohort 3 - Placebo (Placebo Comparator): A single dose of placebo will be administered subcutaneously
  Interventions: Drug: Placebo
- Cohort 4 - Dose 4 of COR-1004 (Experimental): A single dose of COR-1004 will be administered subcutaneously
  Interventions: Drug: COR-1004
- Cohort 4 - Placebo (Placebo Comparator): A single dose of placebo will be administered subcutaneously
  Interventions: Drug: Placebo
- Cohort 5 - Dose 5 of COR-1004 (Experimental): A single dose of COR-1004 will be administered subcutaneously
  Interventions: Drug: COR-1004
- Cohort 5 - Placebo (Placebo Comparator): A single dose of placebo will be administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COR-1004 — COR-1004 administered by subcutaneous (SC) injection
  Arms: Cohort 1 - Dose 1 of COR-1004; Cohort 2 - Dose 2 of COR-1004; Cohort 3 - Dose 3 of COR-1004; Cohort 4 - Dose 4 of COR-1004; Cohort 5 - Dose 5 of COR-1004
Drug: Placebo — Sterile 0.9% (w/v) saline will be used as placebo treatment during the study.
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo; Cohort 5 - Placebo

SUMMARY:
This research study is being done to see if a new, injectable drug called COR-1004 is safe for people to take. It will also help doctors find the right dose of the drug. The study will look at how different dose levels of COR-1004 affect the levels of LDL cholesterol (often called "bad" cholesterol) in the blood. The study will enroll otherwise healthy volunteers who have LDL cholesterol of 100 mg/dl or higher but are not currently taking any cholesterol-lowering medicines.

The main purpose of this study is to test a new drug, COR-1004. Researchers want to find out:

* If the drug is safe and if people have any side effects.
* The highest dose that can be given without causing serious side effects.
* How the body processes the drug.
* How the drug affects the amount of "bad" cholesterol in the blood.

This is an early-phase study. The information learned will help decide if COR-1004 should be tested in larger studies in the future.

To be in this study, you must:

* Be generally healthy.
* Have an LDL ("bad") cholesterol level of 100 mg/dL or higher.
* Not currently be taking any medications to lower your cholesterol.

If you decide to join the study, you will be placed into a group by chance, like flipping a coin. This is called "randomization." In each group, most people (8 out of 10) will get a single injection of the study drug (COR-1004). The other people (2 out of 10) will get a placebo. A placebo looks just like the study drug but has no active medicine in it. Using a placebo helps researchers understand the true effects of the real drug.

This is a "double-blind" study, which means that neither you nor the study doctor will know if you are getting the study drug or the placebo.

The study will test different dose levels of COR-1004. It will start with a low dose and, only if it is proven to be safe, will a new group of participants be given a slightly higher dose. To be extra safe, the first two people in each new dose group will be watched for 24 hours before the other eight people in that group get their injection.

After the injection, you will need to visit the study clinic several times over the next year for follow-up. These visits will include:

* Answering questions about your health.
* Physical exams.
* Blood tests to check your safety and your cholesterol levels.

A special group of experts, called a Safety Review Committee, will carefully watch over the study to protect all participants.

Your active participation in the study, including follow-up visits, will last for about 12 months after you receive the single injection.

Because COR-1004 is a new drug, there may be risks that are not yet known. The study staff will explain all the known risks to you before you agree to participate. Known risks may include discomfort at the injection site, like redness, swelling, or pain. The study team will monitor you very closely for any side effects throughout the study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-ascending-dose study of COR 1004 administered SC to participants with LDL-C ≥100 mg/dL who are otherwise healthy and not on lipid-lowering therapy.

Each cohort will be comprised of 10 participants randomized 4:1 to receive a single dose of study drug or placebo, respectively.

Monitoring will continue on an outpatient basis, with participants returning to the clinical study site for safety, tolerability, PK, PD, and exploratory biomarker monitoring at specified time points through Day 90. Following Day 90, participants will continue to be monitored for adverse events, blood pressure, liver function tests, PD, and exploratory biomarkers through Month 12.

Dosing in Cohorts 1 to 5 will use a sentinel dosing approach, with the first two participants (one active and one placebo) receiving COR-1004 or placebo 24 hours prior to the remainder of the cohort. If deemed safe and tolerated after 24 hours, and no dose-limiting toxicity is observed by the investigator, the remainder of the cohort will be dosed as planned. The sentinel dosing approach will not be utilized for Cohort 6.

ELIGIBILITY:
Inclusion Criteria:

* Serum LDL-C ≥100 mg/dL (≥2.6 mmol/L) at Screening.
* Female participants who are of childbearing potential must be willing to use two highly effective methods of contraception, one of which should be a barrier method.
* Post-menopausal females must be post-menopausal for 12 months.
* Male participants and their partners of child-bearing potential, or same-sex partners, must be willing to use two highly effective methods of contraception, one of which must be a barrier method (eg, condom) for 90 days after study drug administration.
* Able to participate, and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

* Any active or chronic disease.
* Active or history of serious mental illness or psychiatric disorder.
* Clinically significant illness within seven days before study drug administration.
* Having risk of atherosclerotic cardiovascular disease (ASCVD) ≥7.5% based on the ASCVD Risk Estimator Plus.
* Having fasting triglyceride level ≥400 mg/dL (≥4.52 mmol/L).
* Clinically significant abnormalities on physical examination, vital signs, or laboratory test results (except for serum LDL-C) during Screening or prior to admission to the study unit.
* Participants with any risk factors or family history for QT or Fridericia-corrected QT interval (QTcF) prolongation or ECG abnormalities or any abnormality in the ECG.
* Confirmed systolic blood pressure (SBP) >140 mmHg or diastolic blood pressure (DBP) >90 mmHg at Screening, Day -1, or pre-dose.
* Mean resting pulse rate <40 bpm or >90 bpm at Screening.
* Abnormal renal function including serum creatinine greater than the upper limit of normal (ULN) or calculated creatinine clearance <60 mL/min (using the Cockcroft-Gault formula).
* Alanine aminotransferase (ALT) and/or total bilirubin above the ULN. Aspartate aminotransferase (AST), alkaline phosphatase (ALP), or gamma glutamyl transferase (GGT) >2 × ULN. International normalized ratio (INR) above the upper bound of the normal reference range (as per the local laboratory reference range) at Screening.
* Positive hepatitis B surface antigen, hepatitis B virus, hepatitis C virus, or human immunodeficiency virus infection.
* Pregnant or lactating women, or males with female partners who are pregnant or lactating.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide, N-acetylgalactosamine (GalNAc), or inclisiran.
* Participation in an investigational drug or device study within 45 days or five half-lives (whichever time period is longer) or six months for biologic therapies prior to study drug administration.
* Received small interfering ribonucleic acid (siRNA) as an investigational or approved product prior to study drug administration.
* Use of any medications (prescription or over-the-counter) or herbal supplements within two weeks or five half-lives (whichever is longer) prior to study drug administration (six months for biologic therapies), with exception of acetaminophen/paracetamol up to 2 g per day up to 48 hours prior to dosing or medications for contraception. Other exceptions will only be made if the rationale is discussed and clearly documented between the Clinical Research Organization and Sponsor.
* Received any medication, herbal supplements, or nutraceutical known to alter serum lipids within 30 days before Screening (eg, niacin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Clinical and Laboratory Adverse Events within 90 Days post COR-1004 administration | Day 1 to Day 90
  To evaluate the safety and tolerability of COR-1004 when administered subcutaneously as a single dose to otherwise healthy participants with LDL-C ≥100mg/dL
Severity of Clinical and Laboratory Adverse Events within 90 Days post COR-1004 administration | Day 1 to Day 90
  To evaluate the safety and tolerability of COR-1004 when administered subcutaneously as a single dose to otherwise healthy participants with LDL-C ≥100mg/dL

SECONDARY OUTCOMES:
To characterize the maximum observed concentration (Cmax) | Day 1 to Day 90
To characterize the time of maximum observed concentration (Tmax) | Day 1 to Day 90
To characterize the area under the concentration versus time curve (AUC). | Day 1 to Day 90
To characterize the elimination half-life (t1/2). | Day 1 to Day 90
Absolute change from baseline in LDL-C (direct beta quantification method) and PCSK-9 | Day 1 to Day 90
Percent change from baseline in LDL-C (direct beta quantification method) and PCSK-9 | Day 1 to Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes